CLINICAL TRIAL: NCT05222152
Title: A Double-Blind, Double-Dummy, Two-Way Cross-Over, Randomised, Phase II Study of Efficacy, Safety and Tolerability of Modified-Release Hydrocortisones: Chronocort® Versus Plenadren®, in Adrenal Insufficiency
Brief Title: Chronocort Versus Plenadren Replacement Therapy in Adults With Adrenal Insufficiency
Acronym: CHAMPAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIUR-016-AI
Record Dates: First submitted 2021-11-29; First posted 2022-02-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Primary Adrenal Insufficiency
MeSH Terms: conditions — Addison Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chronocort (Experimental): Chronocort (hydrocortisone modified-release hard capsule) supplied as 5 mg and 10 mg strengths will be administered orally. Chronocort 10 mg will be taken on waking (typically between 06:00 and 08:00 hours) and Chronocort 15 mg will be taken just prior to going to bed (typically between 22:00 hours and midnight).
  Interventions: Drug: Chronocort
- Plenadren (Active Comparator): Plenadren (hydrocortisone modified-release tablet) supplied as 5 mg and 20 mg strengths and administered orally. Plenadren 25 mg will be taken on waking (typically between 06:00 and 08:00 hours).
  Interventions: Drug: Plenadren

INTERVENTIONS:
Drug: Chronocort — Hydrocortisone modified-release hard gelatin capsules for oral administration - 5mg and 10mg
  Other Names: Hydrocortisone modified-release hard capsule
  Arms: Chronocort
Drug: Plenadren — Hydrocortisone modified-release tablets for oral administration - 5mg and 20mg
  Other Names: hydrocortisone modified-release tablet
  Arms: Plenadren

SUMMARY:
This study is a double-blind, double-dummy, two-way cross-over, randomised, Phase II study to be conducted at approximately 6 investigational sites in 2 countries. The study will compare the efficacy, safety and tolerability of twice daily Chronocort, a modified-release hydrocortisone, with once daily Plenadren, a modified-release hydrocortisone, over a treatment period of up to 2 months in participants aged 18 years and over, diagnosed with primary Adrenal Insufficiency (AI).

DETAILED DESCRIPTION:
The 4-month study period will comprise a Screening Period of up to 4 weeks (during which participants will receive usual standard of care [SoC] treatment), two 4-week cross-over periods (Treatment Periods 1 and 2), and a 4-week Follow-up Period. Participants will be randomly assigned on a 1:1 basis to either Chronocort in Treatment Period 1 and Plenadren in Treatment Period 2 (Treatment Sequence I), or Plenadren in Treatment Period 1 and Chronocort in Treatment Period 2 (Treatment Sequence II). The total daily dose of Chronocort or Plenadren will be 25 mg according to international guidelines and the Plenadren Summary of Product Characteristics (SmPC). Plenadren 25 mg will be taken once daily in the morning on waking (typically between 06:00 and 08:00 hours). Chronocort 10 mg will be taken in the morning on waking (typically between 06:00 and 08:00 hours) and Chronocort 15 mg will be taken at night just prior to going to bed (typically between 22:00 hours and midnight). Placebo capsules and tablets will be provided to each participant to mask the treatment being received and maintain the study blinding. The first dose of study drug will be taken in the evening of Day 1 and the morning dose on Day 29 will be the last study drug dose in Treatment Period 1. The first dose of study drug in Treatment Period 2 will be taken in the evening of Day 29 and the morning dose on Day 57 will be the last study drug dose in Treatment Period 2 and the end of the dosing periods. The dose will not be changed during the study, but participants will receive stress dosing rules and an emergency treatment pack. Use of stress doses and reasons for use will be collected in an electronic participant diary. If a stress dose is taken within 48 hours before any clinic visit, then the visit should be delayed until the participant has had a 48-hour period without use of any stress doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be aged 18 years or older at the time of signing the informed consent.
* Participants with known (documented) primary AI, defined as early morning pre-dose cortisol <50 nmol/L and currently treated with glucocorticoid as replacement therapy. Primary AI includes any cause of acquired or congenital primary adrenal failure including autoimmune Addison's disease and bilateral adrenalectomy (except when performed for Cushing's syndrome).
* Participants on stable glucocorticoid treatment for ≥3 months prior to the Screening Visit.
* Participants on a stable dose of fludrocortisone (if applicable) for ≥3 months prior to the Screening Visit.
* Male participants must agree to use contraception as detailed in Appendix 4 of the protocol, during the Screening, Treatment, and Follow-up Periods and refrain from donating sperm during these periods and for 7 days after the last dose of study treatment.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and for whom at least one of the following conditions applies: not a woman of childbearing potential (WOCBP), or a WOCBP with a negative urine pregnancy test at entry into the study who agrees to follow the contraceptive guidance during the Screening, Treatment and Follow-up Periods and for 7 days after the last dose of study treatment. Note: Females presenting with oligomenorrhea or amenorrhea who are ≤55 years should be considered potentially fertile (unless permanently sterile) and therefore, as well as undergoing pregnancy testing like all other female participants, will be expected to use an acceptable method of contraception as described in Appendix 4 during the Screening, Treatment and Follow-up Periods and for 7 days after the last dose of study treatment.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.

Exclusion Criteria:

* Participants with Congenital adrenal hyperplasia (CAH).
* Participants with secondary and tertiary AI.
* Past or current history of Cushing's syndrome.
* Adrenal suppression and/or AI induced by exogenous steroids.
* Drug-induced AI.
* Clinical or biochemical evidence of hepatic disease: elevated liver function tests (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >3 times the upper limit of normal [ULN]).
* Clinical or biochemical evidence of renal disease: serum creatinine level of >221 μmol/L (2.5 mg/dL) or calculated creatinine clearance of <25 mL/min.
* History of malignant brain tumours or traumatic brain injury.
* History of malignancy within the last 5 years or treated basal cell carcinoma within the past year.
* Participants who have type 1 diabetes or type 2 diabetes receiving regular insulin.
* Participants with type 2 diabetes whose screening HbA1c exceeds 9%.
* Participants who have elective surgical procedures scheduled during the study.
* Participants with significant medical or psychiatric conditions that in the opinion of the Investigator would preclude participation in the study.
* Participants who have had bariatric surgery within the past 6 months and participants who plan to undertake a major weight loss and/or exercise program during the same time period as anticipated study involvement.
* Restless legs syndrome/Willis-Ekbom disease.
* Participants who have increased gastrointestinal motility e.g., chronic diarrhoea, that may be at risk of impaired cortisol exposure. There are no data in patients with confirmed slow gastric emptying or decreased motility disease/disorder so the clinical response should be monitored in patients with these conditions.
* Participants anticipating regular prophylactic use of additional steroids e.g., for strenuous exercise.
* Participants with co-morbidities requiring daily administration of a medication (or consumption of any material) that interferes with the metabolism of glucocorticoids.
* Participants on regular daily inhaled, topical, nasal, or oral steroids for any indication other than AI.
* Participants who have received intra-articular steroid injections within 1 year prior to the Screening Visit or for whom such injections are planned during the study.
* Participants who are receiving <10 mg hydrocortisone dose at the Screening Visit or the hydrocortisone dose equivalent.
* Participants taking sleeping medication.
* Participants treated at screening with either Chronocort or Plenadren.
* Participation in another clinical study of an investigational or licensed drug or device within 12 weeks or 5 half-lives prior to the Screening Visit or at any time during study participation.
* Active alcohol or drug abuse within 1 year prior to the Screening Visit.
* Participants who routinely work night shifts and do not sleep during the usual night-time hours.
* Participants who intend to travel and cross a time zone of greater than ±3 hours within 1 week of the scheduled visit dates.
* Participants unable to comply with the requirements of the protocol in the opinion of the Investigator.
* Participants with a known hypersensitivity to any of the components of the Chronocort capsules, the Plenadren tablets, the Chronocort placebo, or the Plenadren placebo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
To measure the change in morning serum cortisol levels from baseline, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  The primary efficacy outcome variable is the 07:00 hour serum cortisol level after 4 weeks of treatment. The treatment effect (Chronocort minus Plenadren, after logarithmic transformation) will be estimated in the efficacy evaluable analysis set (EEAS) (defined as participants with morning serum cortisol assessed at baseline and after each treatment period, with no major protocol violations) using a linear mixed model.

SECONDARY OUTCOMES:
To measure change in morning fatigue from baseline, using the Multidimensional Assessment of Fatigue (MAF) questionnaire within 1 hr of waking, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  MAF morning fatigue score after 4 weeks of treatment. MAF is a 16 item scale that measures fatigue according to 4 dimensions; degree and severity, distress that it causes, timing of fatigue, and it's impact of various activities of daily living to give a Global Fatigue Score of up to 50, where a higher value equates to more fatigue.
To measure the change from baseline, in terms of achieving physiological morning cortisol levels after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  Whether or not a participant has achieved a physiological morning cortisol level (defined as the 07:00 hour serum cortisol before the morning dose of >140 nmol/L after 4 weeks of treatment) will be summarised and compared between treatment periods.
  Note: a morning cortisol level below 140 nmol/L is considered to reflect relative AI in international guidelines [Bornstein, 2016].
To measure the change from baseline in terms of closeness of overall salivary cortisone levels during the day to a normal physiological profile, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  A salivary cortisone profile score will be derived at the end of 4 weeks of treatment. The profile score is calculated by comparing the on-study salivary cortisol profile with a profile obtained from healthy volunteers. Five timepoints are compared, where a more similar profile to the normal healthy volunteer profile is preferred.
To measure the change from baseline in ACTH control in the morning, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  The 07:00 hour plasma ACTH level after 4 weeks of treatment will be summarised and compared between treatment periods.
To measure the change from baseline to the bone marker of osteocalcin, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  Osteocalcin levels after 4 weeks of treatment will be summarised and compared between treatment periods.
To measure the change from baseline in morning fatigue using the PROMIS® 7b questionnaire within 1 hour of waking, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  Morning fatigue, using the Patient-Reported Outcomes Measurement Information System (PROMIS® 7b) questionnaire, within 1 hour of waking after 4 weeks of treatment will be summarized and compared between treatment periods. PROMIS 7b is a 7-item scale that measures self-reported fatigue that may impact daily activities and normal functioning. A higher PROMIS 7b score indicates greater fatigue and therefore a less favorable outcome.
To measure the change from baseline in QoL using the EuroQol 5-level Standardized Health Questionnaire (EQ-5D-5L™), after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  QoL, using the EQ-5D-5L after 4 weeks of treatment, will be summarized and compared between treatment periods. The scale measures on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Where the minimum score is 0 and maximum score is 100, a high score indicates a more favorable outcome.
To measure the change from baseline in QoL using the Health-related Quality of Life in Addison's disease (AddiQoL) questionnaire, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  QoL, using the AddiQoL questionnaire after 4 weeks of treatment, will be summarized and compared between treatment periods. AddiQoL is a 30 item scale measuring health-related quality of life in Addison's disease. A higher score indicates a higher quality of life and therefore a more favorable outcome.
To measure the change from baseline in terms of QoL using the 36-Item Short Form Health Survey (SF-36®) questionnaire, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  QoL, using SF-36 questionnaire after 4 weeks of treatment, will be summarized and compared between treatment periods. Analyses of SF-36 at other timepoints are exploratory analyses. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). All components contribute in different proportions to the overall measures. Where the minimum score is 0 and maximum score is 100 and a high score is a more favorable score.

OTHER OUTCOMES:
To measure the change in terms of activity, after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | After the end of each 4 week treatment period.
  Mean daily steps, mean steps between 07:00-15:00 hours, and mean steps between 15:00-23:00 hours, as assessed by a wearable device, will be summarized and compared between treatment periods, where more steps, i.e. more activity is considered preferable.
To measure the change in terms of sleep, after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | After the end of each 4 week treatment period.
  Mean sleep hours, mean rapid eye movement (REM) sleep, mean light sleep, and mean deep sleep, as assessed by a wearable device, will be summarized and compared between treatment periods, where greater length of sleep is considered preferable.
To measure the change from baseline in terms of QoL using the Diurnal Alertness visual analogue scale (VAS), after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  QoL, using the Diurnal Alertness VAS, after 4 weeks of treatment and at other timepoints will be summarized and compared between treatment periods. QoL will be assessed using a Visual Analog Scale (VAS), which is a 10cm scale ranging from 'Brain Fog: unable to perform normal daily tasks' to 'Fully Alert: able to perform normal daily tasks easily'. A higher score indicates a better outcome.
To measure the change from baseline in terms of QoL using the General Anxiety Disorder-7 (GAD-7) scale, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  The GAD-7 scale is a screening tool and symptom severity measure for the seven most common anxiety disorders. QOL measured using the GAD-7 scale after 4 weeks of treatment and at other timepoints will be summarized and compared between treatment periods. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions, where a lower score indicates a better outcome.
To measure the change from baseline in terms of QoL using the Patient Health Questionnaire-9 (PHQ-9) scale, after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  The PHQ-9 is a self-administered assessment scale for the evaluation of depression symptoms. QoL, using the PHQ-9 scale, after 4 weeks of treatment and at other timepoints will be summarized and compared between treatment periods. The PHQ-9 scale consists of 9 questions, each with a score of 0-3, with 0 meaning Not at All, 1 meaning Several Days, 2 meaning More than half of the days and 3 Nearly every day. As the score increases then this is indicative of a more serious depressive disorder. There is a 10th question which is only answered if one of the scores for questions 1 to 9 are 1 or more.
To measure the change from baseline in terms of QoL using the Gissen Complaints Questionnaire-24 (GBB-24) scale (German participants only), after 4 weeks treatment with Chronocort compared with 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  The GBB-24 scale measures self reported physical complaints in terms of whether the issue is fully or partially psychosomatically induced. QoL, using the GBB-24 scale, after 4 weeks of treatment and at other timepoints will be summarized and compared between treatment periods. The GBB-24 consists of 24 different health complaints, the severity of each is rated according to a five point scale; 0 (not at all), 1 (slightly), 2 (somewhat), 3 (considerably) and 4 (very much) [23]. The complaints are grouped and summarized into four subscales with six complaints in each of the following groups: Cardiovascular complaints, gastrointestinal complaints, musculoskeletal complaints and exhaustion, where a lower score indicates a more favorable outcome.
To assess the participant's preference to treatment, after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | After the end of each 4 week treatment period.
  Participant preference for assigned treatment during Treatment Period 1 relative to pre-study treatment, and for assigned treatment during Treatment Period 2 relative to that during Treatment Period 1, will be summarised and compared between treatments.
To assess treatment compliance, after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | After the end of each 4 week treatment period.
  The percentage treatment compliance between visits and overall will be summarised.
To measure change in terms of safety and tolerability, after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | After the end of each 4 week treatment period.
  The incidence, nature, severity, relatedness, duration, outcome, seriousness, and expectedness of treatment-emergent adverse events (TEAEs) will be tabulated by treatment period.
To measure change from baseline in terms of blood pressure, after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  Blood pressure after 4 weeks of treatment will be summarised and compared between treatment periods.
To measure change from baseline in terms of glycated haemoglobin (HbA1c), after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  HbA1c levels after 4 weeks of treatment will be summarised and compared between treatment periods.
To measure the change in terms of stress dosing (use of participant administered emergency treatment pack), after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | After the end of each 4 week treatment period.
  The number of extra doses per period will be summarised and compared between treatment periods.
To measure the change from baseline in terms of lipid profile, after 4 weeks treatment with Chronocort compared to 4 weeks treatment with Plenadren (crossover study). | Baseline and end of each 4 week treatment period.
  Total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, very low density lipoprotein (VLDL) cholesterol, triglycerides, apolipoprotein (Apo) A-I, Apo B, and lipoprotein(a) (Lp(a)) will be summarized and compared between treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: R Ross, Principal Investigator — Neurocrine UK Limited
Locations (7):
- Germany (3):
  - Diurnal Investigational Site in Hamburg, Hamburg
  - Diurnal Investigational Site in Munich, Munich
  - Diurnal Investigational Site in Würzburg, Würzburg
- United Kingdom (4):
  - Diurnal Investigational Site in Birmingham, Birmingham
  - Diurnal Investigational Site in Cardiff, Cardiff
  - Diurnal Investigational Site in Newcastle, Newcastle
  - Diurnal Investigational Site in Sheffield, Sheffield

REFERENCES:
- [Derived] Prete A, Theiler-Schwetz V, Arlt W, Hazeldine J, Chifu IO, Harbeck B, Napier C, Newell-Price JDC, Rees DA, Reisch N, Stalla GK, Coope H, Maltby K, Porter J, Quirke J, Ross RJ. Effects of modified release hydrocortisone on restoration of early morning cortisol, quality of life, and fatigue in adrenal insufficiency (The CHAMPAIN study): a randomised, double-blind, double-dummy, cross-over study comparing Chronocort and Plenadren. EClinicalMedicine. 2026 Jan 2;91:103714. doi: 10.1016/j.eclinm.2025.103714. eCollection 2026 Jan. PMID 41552007